CLINICAL TRIAL: NCT01170780
Title: Dexamethasone Versus Placebo in Optimizing the Postoperative Period After Laparoscopic Inguinal Hernia Repair
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mette Astrup Madsen (Other)
Responsible Party: Sponsor-Investigator, Mette Astrup Madsen, M.D., Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: dx3
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Inguinal Hernia; Femoral Hernia
Keywords: Inguinal hernia; Transabdominal preperitoneal hernia repair; TAPP; Dexamethasone; Pain
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Femoral; Pain | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Saline
- Dexamethasone (Active Comparator): Corticosteroid (Fortecontin 8 mg)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — single use of dexamethasone IV 8 mg/2 ml
  Other Names: Fortecontin
  Arms: Dexamethasone
Drug: Saline — 2 ml IV
  Other Names: Natriumchlorid, B. Braun 9 mg/ml
  Arms: Placebo

SUMMARY:
Does corticosteroid (dexamethasone) have an effect on the postoperative period after laparoscopic hernia repair, when it comes to pain, postoperative nausea and vomiting and convalescence. This randomized, double-blinded study compares dexamethasone versus placebo. The patients are recommended one day of convalescence. The medicine or placebo is given before operation. The patients fill out questionnaire before operation and three hours after operation and in the following three days. The patients also register when they return to normal activities and work.

ELIGIBILITY:
Inclusion Criteria:

* patients planned for elective laparoscopic hernia repair (TAPP)
* Unilateral inguinal or femoral hernia
* ASA class I-II
* Read and speak Danish

Exclusion Criteria:

* Acute hernia operation
* Operation for other hernias with mesh during the same procedure
* Endocrine disease (diabetes, adrenal insufficiency etc.)
* fever/infection within the first 10 days before operation
* Poor compliance
* No signed consent form
* Daily intake of opioids or anxiolytic drugs
* Manic episodes
* Use medicine against glaucoma
* Use thiazide or loop diuretics
* Vaccination within the last 14 days

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
pain during coughing | day 1
  Assessed with visual analog scale (VAS 0-100 mm)

SECONDARY OUTCOMES:
pain during coughing | 4 days
  Assessed with VAS
pain at rest | 4 days
  Assessed with VAS
convalescence | 1 month
  Registration of number of days after operation before returning to work and recreational activities.
pain at rest | 4 days
  Assessed with verbal rating scale (VRS:no pain, mild pain, severe pain, worst thinkable pain)
nausea | 2 days
  Assessed with verbal rating scale (VRS: no nausea, mild nausea, severe nausea, worst thinkable nausea)
vomiting | 2 days
  yes/no question. If yes, how many times have you been vomiting?
discomfort | 4 days
  Assessed with visual analog scale (VAS, 0-100 mm)
fatigue | 4 days
  Assessed with numeric rating scale (NRS, 1-10)

CONTACTS AND LOCATIONS:
Overall Officials: Mette A Tolver, M.D., Principal Investigator — University Hospital Koege; Thue Bisgaard, M.D. DMSc, Principal Investigator — University Hospital Koege
Locations (1):
- University Hospital Koege, Koege, Denmark

REFERENCES:
- [Derived] Tolver MA, Strandfelt P, Bryld EB, Rosenberg J, Bisgaard T. Randomized clinical trial of dexamethasone versus placebo in laparoscopic inguinal hernia repair. Br J Surg. 2012 Oct;99(10):1374-80. doi: 10.1002/bjs.8876. PMID 22961516